CLINICAL TRIAL: NCT04034342
Title: The Effect of RaceRunning on Cardiometabolic Disease Risk Factors and Functional Mobility in Young People With Moderate-to-severe Cerebral Palsy: a Feasibility Study
Brief Title: RaceRunning for Young People With Moderate-to-severe Cerebral Palsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Queen Margaret University (Other)
Collaborators: Brunel University (Other); University of Gloucestershire (Other); University of Edinburgh (Other)
Responsible Party: Principal Investigator, Marietta van der Linden, Senior Research Fellow, Queen Margaret University
Other Study IDs: 259279
Record Dates: First submitted 2019-07-15; First posted 2019-07-26 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Exercise; Cerebral Palsy
Keywords: RaceRunning;; cardiometabolic health desease risk; functional mobility
MeSH Terms: conditions — Motor Activity; Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: RaceRunning — RaceRunning (www.racerunning.org) is a growing disability sport that provides an opportunity for people with moderate-to-severe CP to participate in exercise in the community. It allows those who are unable to walk independently, to propel themselves using a RaceRunning bike, which has a breastplate for support but no pedals. Participants sit on the saddle and use their legs to propel themselves forward.

SUMMARY:
Physical inactivity in people with cerebral palsy (CP) has been linked with increased risk of cardiometabolic disease. Exercise studies rarely include people with CP with severe walking impairments and assess the sustainability of the intervention. RaceRunning allows people severe walking impairments to independently propel themselves using a running bike, which has a breast plate for support but no pedals. This project will assess the feasibility of at trial into the effectiveness of RaceRunning to reduce cardiometabolic disease risk factors and improve functional mobility. Intervention: Weekly standardised RaceRunning sessions over 6 months led by an experienced coach. Participants Twenty-five young people with CP aged 5-21, GMFCS levels III-V. Feasibility outcomes: Acceptability of RaceRunning, adherence and fidelity of the intervention, recruitment and retention rates and adverse events. Outcome measures: Cardiometabolic disease risk factors (physical activity, sedentary time, resting heart rate and blood pressure and aerobic capacity) and functional mobility assessed at baseline, 3 and 6 months. Quality of life (EQ-5D-Y) and health service use will inform a future cost-effectiveness analysis. Aspects of feasibility and acceptability and the variability and patterns of the change in outcomes will be reported using descriptive statistics.

DETAILED DESCRIPTION:
This is a multi-centre experimental study with a single intervention arm. Assessments will be conducted at baseline, 12 weeks and 24 weeks. The intervention will be delivered in Scotland and Gloucestershire. Participants will take part in one RaceRunning session each week for a period of 24 weeks. The content of the sessions will be standardised for all training groups and will consist of a warm-up, coordination (drills), sprint and endurance training, and cool-down. The training program will be adapted to the athlete's ability and fitness. The project objectives are to examine the feasibility of delivering and acceptability of participating in RaceRunning as a community-based intervention for young people with moderate-to-severe CP, including fidelity to and safety of the intervention. Secondly, to examine the feasibility of conducting a definitive study of RaceRunning including exploring recruitment and retention over 24 weeks, acceptability of data collection methods and rate of outcome measure completion, and acceptability and quantity of missing data relating to health economic data collection tools. Finally, to examine the variability and patterns of change in outcomes over 24 weeks in order to determine a primary outcome measure and calculate sample size for a future study.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of cerebral palsy or brain injury affecting coordination
* Aged 5 to 21
* GMFCS E-R level III, IV or V
* Less than 15 hours of RaceRunning experience
* Able to independently propel the bike for at least 30 meters
* An ability to comprehend and follow instructions relating to participation in RaceRunning training

Exclusion Criteria:

* Lower limb surgery
* Having started Botox or other spasticity treatment less than 6 months prior to the start of the study
* Severe visual impairment affecting the ability to safely take part in RaceRunning training sessions

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: It is envisaged that the cohort will be recruited from a variety of RaceRunning clubs in Scotland: Meadowmill RaceRunning squad, Pitreavie AC (Dumfermline), if required Perth AC, Forth Valley Flyers, Ayr Seaforth AC and Glasgow Victoria Park AC. The participants in England will be recruited from Gloucester athletics club and Milestones school.
  The RaceRunning clubs and the study will be advertised through appropriate social media channels (Facebook, Twitter) and websites such as Scottish Disability Sport, Cerebral Palsy Scotland, CP Sport England etc. to further increase the recruitment potential.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
maximum aerobic capacity (VO2max) | Baseline, 12 weeks and 24 weeks
  an incremental test protocol will be used to measure the maximum oxygen uptake (ml/ min kg) an incremental test protocol will be used to measure maximum oxygen uptake (ml/min kg)

SECONDARY OUTCOMES:
Physical activity | Baseline, 12 weeks and 24 weeks
  The number of steps over five 24 hour periods will be recorded using an activity monitor.
sedentary behaviour | Baseline, 12 weeks and 24 weeks
  The time (in minutes) spent in an lying or sitting over five 24 hour periods will recorded using an activity monitor.
Resting heart rate (beats per min) | Baseline, 12 weeks and 24 weeks
  The average heart rate during 2 minutes of quiet sitting
Resting heart rate blood pressure (mmHg) | Baseline, 12 weeks and 24 weeks
  The average blood pressure during 2 minutes of quiet sitting
Functional mobility Scale | Baseline, 12 weeks and 24 weeks
  The Functional Mobility Scale (FMS) will be used to describe the level of a child's mobility in everyday life over 5m, 50m, and 500m and representing the home, school and community settings respectively.
Muscle strength | Baseline, 12 weeks and 24 weeks
  Knee extensor strength (N) will be assessed with a hand-held dynamometry
calf and waist circumference (mm) | Baseline, 12 weeks and 24 weeks
  The circumference of the calf and waist will be measured using a tape measure
Quality of Life (EQ-5D) | Baseline, 12 weeks and 24 weeks
  The EQ-5D-Y/EQ-5D-5L will be used to describe and value the health in terms of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
The Canadian Occupational Performance Measure | Baseline, 12 weeks and 24 weeks
  The Canadian Occupational Performance Measure will be used to identify important activities for each participant and to record the change in participants' perceived performance rating of this activity and the satisfaction of this performance over time. psychosocial outcomes such as happiness, self-esteem, independence and quality of life.
Psychosocial Impact of Assistive Devices Scale (PIADS) | Baseline, 12 weeks and 24 weeks
  The PIADS will be used to record the change in psychosocial outcomes such as happiness, self-esteem, independence and quality of life as a result of using a specific assistive device (RaceRunner).

CONTACTS AND LOCATIONS:
Overall Officials: Marietta L van der Linden, PhD, Principal Investigator — Queen Margaret University
Locations (2):
- United Kingdom (2):
  - University of Gloucestershire, Gloucester
  - Queen Margaret University, Musselburgh

REFERENCES:
- [Derived] Ryan J, Theis N, Koufaki P, Phillips S, Anokye N, Andreopoulou G, Kennedy F, Jagadamma KC, vanSchie P, Dines H, van der Linden ML. Effect of RaceRunning on cardiometabolic disease risk factors and functional mobility in young people with moderate-to-severe cerebral palsy: protocol for a feasibility study. BMJ Open. 2020 Jul 1;10(7):e036469. doi: 10.1136/bmjopen-2019-036469. PMID 32611743